CLINICAL TRIAL: NCT06641817
Title: An Observed Research: to Assess Kawasaki Disease with Cardiovascular Imaging
Brief Title: The Value of Cardiovascular Imaging in Kawasaki Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: West China Second University Hospital (Other)
Responsible Party: Principal Investigator, Ling-Yi Wen, Principal Investigator, West China Second University Hospital
Other Study IDs: WestChinaSUH2023095-2
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Kawasaki Disease
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The whole boold including blood cell and plasma will be collected for laboratory and genetic test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- petients diagnosed with Kawasaki disease: Diagnostic criteria: based on the American Heart Association(AHA) guideline

SUMMARY:
The goal of this observational study is to assess the cardiovascular injury of Kawasaki disease with multi-modal imaging combined with clinical data.

During their disease progress, participants will undergo cardiovascular magnetic resonance, echocardiography, electrocardiography, laboratory tests, and genetic tests when hospitalization and follow-up, and the baseline data will be collected at the admission. Some patients will undergo coronary computed tomography angiography (CCTA) or DSA due to the disease progress. All the above examination data and changes will be analyzed to assess the value of cardiovascular imaging in the pathogenesis, diagnosis, and prognosis of Kawasaki disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed based on the American Heart Association guideline for Kawasaki disease.

Exclusion Criteria:

* Patients with a history of congenital heart disease, cardiomyopathy.
* Patients with age over 18 years old.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: From the past to Jaunary 2033, pediatric patients diagnosed with Kawasaki disease were recruited from West China Second University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2033-01-01 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 10 years after the onset
  Major adverse cardiovascular events including cardiac death, transient ischemic attack or stroke, myocardial infarction, arrhythmia, heart failure, severe valvular disease, percutaneous coronary intervention, coronary artery bypass graft, and other cardiovascular surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University., Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kuroda H, Oguri T, Kamiyama N, Toyoda H, Yasuda S, Imajo K, Suzuki Y, Sugimoto K, Akita T, Tanaka J, Yasui Y, Kurosaki M, Izumi N, Nakajima A, Fujiwara Y, Abe T, Kakisaka K, Matsumoto T, Kumada T. Multivariable Quantitative US Parameters for Assessing Hepatic Steatosis. Radiology. 2023 Oct;309(1):e230341. doi: 10.1148/radiol.230341. PMID 37787670
- [Background] Xie LP, Yan WL, Huang M, Huang MR, Chen S, Huang GY, Liu F. Epidemiologic Features of Kawasaki Disease in Shanghai From 2013 Through 2017. J Epidemiol. 2020 Oct 5;30(10):429-435. doi: 10.2188/jea.JE20190065. Epub 2019 Sep 21. PMID 31548437
- [Background] Chen JJ, Ma XJ, Liu F, Yan WL, Huang MR, Huang M, Huang GY; Shanghai Kawasaki Disease Research Group. Epidemiologic Features of Kawasaki Disease in Shanghai From 2008 Through 2012. Pediatr Infect Dis J. 2016 Jan;35(1):7-12. doi: 10.1097/INF.0000000000000914. PMID 26372452
- [Background] Vranicar M, Hirsch R, Canter CE, Balzer DT. Selective coronary angiography in pediatric patients. Pediatr Cardiol. 2000 May-Jun;21(3):285-8. doi: 10.1007/s002460010064. PMID 10818198
- [Background] Suda K, Iemura M, Nishiono H, Teramachi Y, Koteda Y, Kishimoto S, Kudo Y, Itoh S, Ishii H, Ueno T, Tashiro T, Nobuyoshi M, Kato H, Matsuishi T. Long-term prognosis of patients with Kawasaki disease complicated by giant coronary aneurysms: a single-institution experience. Circulation. 2011 May 3;123(17):1836-42. doi: 10.1161/CIRCULATIONAHA.110.978213. Epub 2011 Apr 18. PMID 21502578
- [Background] McCrindle BW, Rowley AH, Newburger JW, Burns JC, Bolger AF, Gewitz M, Baker AL, Jackson MA, Takahashi M, Shah PB, Kobayashi T, Wu MH, Saji TT, Pahl E; American Heart Association Rheumatic Fever, Endocarditis, and Kawasaki Disease Committee of the Council on Cardiovascular Disease in the Young; Council on Cardiovascular and Stroke Nursing; Council on Cardiovascular Surgery and Anesthesia; and Council on Epidemiology and Prevention. Diagnosis, Treatment, and Long-Term Management of Kawasaki Disease: A Scientific Statement for Health Professionals From the American Heart Association. Circulation. 2017 Apr 25;135(17):e927-e999. doi: 10.1161/CIR.0000000000000484. Epub 2017 Mar 29. PMID 28356445